CLINICAL TRIAL: NCT05085756
Title: Swedish Partnership in the WHO-WMH-ICS Study on National Mapping and E-health Interventions for Mental Health Issues Among University Students: Psychological Internet Treatment for Improved Mental Health
Brief Title: Transdiagnostic Internet Intervention to Improve Mental Health Among University Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Linkoeping University (Other Government); Malmö University (Other); Stockholm University (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-03599
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Psychological Disorder
MeSH Terms: conditions — Mental Disorders | interventions — bbc3 protein, zebrafish

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided treatment (Active Comparator): 8-week transdiagnostic CBT with written guidance from M.Sc-level students under supervision.
  Interventions: Behavioral: Puma
- Unguided treatment (Active Comparator): 8-week transdiagnostic CBT without guidance.
  Interventions: Behavioral: Puma
- Waitlist (Other): 8-week transdiagnostic CBT without guidance, made available 6 months after recruitment.
  Interventions: Behavioral: Puma

INTERVENTIONS:
Behavioral: Puma — One psychoeducation module followed by two transdiagnostic modules tailored to primary depression or anxiety symptoms, followed by three participant-choice modules, and ending with two transdiagnostic modules.

SUMMARY:
This study offers transdiagnostic CBT-based treatment for symptoms of depression and anxiety to university students who have previously responded to the WHO-WMH-ICS survey.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 cutoff for mild depression
* GAD-7 cutoff for mild anxiety

Exclusion Criteria:

* Suicidal ideation or plans
* Severe levels of mental ill-health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 for depression | last 2 weeks
  9 items measuring depressive symptoms
GAD-7 for anxiety | last 2 weeks
  7 items measuring anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Dept of Psychology, Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
This is a future plan. Outcome data will be shared as appropriate, but primarily within the WHO-WMH-ICS consortium.

REFERENCES:
- [Background] Andersson C, Bendtsen M, Lindfors P, Molander O, Lindner P, Topooco N, Engstrom K, Berman AH. Does the management of personal integrity information lead to differing participation rates and response patterns in mental health surveys with young adults? A three-armed methodological experiment. Int J Methods Psychiatr Res. 2021 Dec;30(4):e1891. doi: 10.1002/mpr.1891. Epub 2021 Aug 21. PMID 34418224
- [Background] Berman AH, Topooco N, Lindfors P, Bendtsen M, Lindner P, Molander O, Kraepelien M, Sundstrom C, Talebizadeh N, Engstrom K, Vlaescu G, Andersson G, Andersson C. Transdiagnostic and tailored internet intervention to improve mental health among university students: Research protocol for a randomized controlled trial. Trials. 2024 Mar 1;25(1):158. doi: 10.1186/s13063-024-07986-1. PMID 38429834